CLINICAL TRIAL: NCT03206086
Title: Eltrombopag for Patients With Fanconi Anemia
Brief Title: Eltrombopag for People With Fanconi Anemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 170121; 17-H-0121
Record Dates: First submitted 2017-06-30; First posted 2017-07-02 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08-21

CONDITIONS: Fanconi Anemia
Keywords: DNA Repair; Inflammation; Hematopoiesis; Pancytopenia
MeSH Terms: conditions — Fanconi Anemia; Inflammation; Pancytopenia | interventions — eltrombopag

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Group (Experimental): Eltrombopag
  Interventions: Drug: Eltrombopag

INTERVENTIONS:
Drug: Eltrombopag — Daily dose - Non-Asian (>=12): 150 mg Non-Asian (6-11): 75 mg East Asian, South East Asian (>=12): 75 mg East Asian, South East Asian (6-11): 37.5 mg

SUMMARY:
Background:

Fanconi anemia is a genetic disease. Some people with it have reduced blood cell counts. This means their bone marrow no longer works properly. These people may need blood transfusions for anemia (low red blood cells) or low platelet counts or bleeding. Researchers want to see if a new drug will help people with this disease.

Objective:

To find out if a new drug, eltrombopag, is effective in people with Fanconi anemia. To know how long the drug needs to be given to improve blood counts.

Eligibility:

People at least 6 years old with Fanconi anemia with reduced blood cell counts.

Design:

Participants will be screened with blood and urine tests. They will repeat this before starting to take the study drug.

Participants will take eltrombopag pills by mouth once a day for 24 weeks. They will be monitored closely for side effects.

Participants will have blood tests every 2 weeks while on eltrombopag.

Participants will visit NIH 3 months and 6 months after starting eltrombopag. At these visits, participants will:

Answer questions about their medical history, how they are feeling, and their quality of life

Have a physical exam

Have blood and urine tests

Have a bone marrow sample taken by needle from the hip. The area will be numbed.

If participants blood cell counts improve, they might join the extended access part of the study. They will continue taking eltrombopag for 3 years and sign a different consent.

After 24 weeks of treatment, if there is no improvement in blood cell counts, participants will stop taking eltrombopag. They will return for an optional follow-up visit that repeats the study visits....

DETAILED DESCRIPTION:
Fanconi anemia (FA) is a rare genetic disease that often presents as a bone marrow failure (BMF) syndrome but also can affect any other organ. Etiologically, loss of function mutations in more than 21 different gene members of the FA core complex (i.e. FANCA-FANCV) have been associated with FA. The FA core complex is involved in interstrand cross-link DNA damage repair during cell division. Impaired DNA repair causes genomic instability which consequently can cause apoptosis of the cell or malignant transformation. In addition to impaired DNA repair mechanisms, FA cells exhibit increased sensitivity to pro-inflammatory cytokines (e.g. IFN-gamma, TNF-alpha) and elevated levels of these cytokines have been associated with bone marrow failure in subjects with FA and other inherited bone marrow failure syndromes.

Patients with FA may present with congenital anomalies, such as microcephaly or short stature. However, the failure of the hematopoietic stem cell (HSC) compartment to produce sufficient numbers of peripheral blood cells, and progression to myelodysplastic syndrome (MDS) and acute myelogenous leukemia (AML) are the greatest risk factors for morbidity and mortality, particular in young patients with FA. In a few reported cases, spontaneous somatic reversion of inherited mutations has resulted in a selective growth advantage of corrected HSCs that subsequently restored hematopoiesis. However, therapeutic options are limited in FA. Although HSC transplantation outcomes have significantly improved over the past two decades, donor availability, graft failure, and FA-specific transplant toxicities are still significant hurdles towards a curative treatment of FA-associated BMF. Moreover, attempts at genetic correction of FA are not yet ready for patient care.

The thrombopoietin (TPO) mimetic eltrombopag (EPAG) has recently been shown to be effective in restoring tri-lineage hematopoiesis in patients with treatment refractory acquired severe aplastic anemia (SAA). Of particular interest for patients with FA is the observation that EPAG also improves the repair of double strand DNA breaks, a mechanism that is impaired in patients with FA. Additionally, our pre-clinical studies indicate that EPAG evades INF-gamma blockade of signal transduction from the TPO receptor (cMPL) resulting in improved survival and proliferation of HSCs. Based on these clinical and pre-clinical studies, we hypothesize that EPAG will improve peripheral blood cell counts in patients with FA and thus reduce morbidity and mortality.

This phase II clinical trial proposes to treat patients with FA for 6 months with EPAG to assess safety and efficacy at improving hematological manifestations of FA. Responders at 6 months will be able to continue EPAG on the extension part of this protocol for an additional 3 years. During this time frame we anticipate further improvement of peripheral blood cells counts that will eventually result in the discontinuation of EPAG after a tapering period. Translational studies will explore EPAG effects on DNA repair activity, apoptosis, global transcriptome and TPO signaling pathways in patient s hematopoietic stem and progenitor cells (HSPCs).

ELIGIBILITY:
* INCLUSION CRITERIA:
* Confirmed diagnosis of Fanconi anemia. Diagnosis is confirmed by a biallelic mutation in a known FANC gene and/or by positive chromosome breakage analysis in lymphocytes and/or skin fibroblasts (for mosaicism).
* One or more of the following three clinically-significant cytopenias: platelet count <= 50,000/microliter or platelet-transfusion-dependence (requiring at least 4 platelet transfusions in the 8 weeks prior to study entry, see definition of platelet transfusion units at 8.2.1); neutrophil count less than 1000/microliter; hemoglobin less than 10 g/dL or red cell transfusion- dependence (requiring at least 4 transfusions of PRBCs (adult patient 4 units PRBC, pediatric patients at least 10ml/kg/transfusion) in the eight weeks prior to study entry.
* Failed or declined treatment with androgens (danazol or oxymetholone).
* Age >= 6 years old.
* Weight >=10kg.

EXCLUSION CRITERIA:

* Known active or uncontrolled infections not adequately responding to appropriate therapy.
* Evidence for MDS or AML as defined by WHO criteria.
* Any cytogenetic abnormality associated with poor prognosis in FA, including gains of chromosome 3q, gains of chromosome 1q, deletions of chromosome 7, and complex cytogenetics (88-90) identified from bone marrow aspirate. Patients with known biallelic mutations in BRCA2 (FANCD1).
* Active malignancy or likelihood of recurrence of malignancies within 12 months
* Moribund status such that death within 7 to 10 days is likely. Comorbidities of such severity that in the view of the investigator it would likely preclude the patient's ability to tolerate eltrombopag.
* Treatment with androgens (danazol or oxymetholone) less than 4 weeks prior to initiating eltrombopag.
* Creatinine > 2.5 times ULN
* Direct Bilirubin > 3.0mg/dL, indicating congenital abnormalities in the bilirubin level
* SGOT (AST) or SGPT (ALT) >5 times the ULN normal
* Known liver cirrhosis in severity that would preclude tolerability of eltrombopag as evidenced by albumin < 35g/L
* Known immediate or delayed hypersensitivity to EPAG or its components
* Female subjects who are nursing or pregnant (positive serum or urine Beta-human chorionic gonadotrophin (Beta-hCG pregnancy test) at screening or pre-dose on Day 1.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for 30 days after the last dose of EPAG. Highly effective contraception methods include:

  * Total abstinence (when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
  * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
  * Male sterilization (at least 6 months prior to screening). For female patients on the study the vasectomized male partner should be the sole partner for that patient.
  * Use of oral, injected or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS), or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception.
  * In case of use of oral contraception women should have been stable on the same pill for a minimum of 3 months before taking study treatment.
  * Women are considered post-menopausal and not of child bearing potential if they have had over 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile age appropriate (e.g. generally 40-59 years), history of vasomotor symptoms (e.g. hot flushes) in the absence of other medical justification or have had surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of childbearing potential.
  * Sexually active males unless they use a condom during intercourse while taking the study treatment and for 30 days after stopping study treatment and should not father a child in this period. A condom is required to be used also by vasectomized men as well as during intercourse with a male partner in order to prevent delivery of the drug via seminal fluid.
* History of thromboembolic events.
* Unable to take oral medication
* History or current diagnosis of cardiac disease indicating significant risk of safety for patients participating in the study such as uncontrolled or significant cardiac disease, including any of the following:

  * Recent myocardial infarction (within last 6 months),
  * Uncontrolled congestive heart failure,
  * Unstable angina (within last 6 months)
  * Clinically significant (symptomatic) cardiac arrhythmias (e.g., sustained ventricular tachycardia, and clinically significant second or third-degree AV block without a pacemaker.)
  * Long QT syndrome, family history of idiopathic sudden death, congenital long QT syndrome or additional risk factors for cardiac repolarization abnormality, as determined by the investigator.
  * Impaired cardiac function such as corrected QTc>450msec using Fridericia correction on the screening EKG, other clinically significant cardio-vascular diseases (e.g. uncontrolled hypertension, history of labile hypertension), history of known structural abnormalities (e.g. cardiomyopathy).
* History of HIV positivity.
* History of alcohol/drug abuse.
* Concurrent participation in an investigational study within 30 days prior to enrollment or within 5-half-lives of the investigational product, whichever is longer. Note: parallel enrollment in a disease registry is permitted.

Ages: 6 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-11-02 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of drug responders | 6 months
  Peripheral blood platelet count increases to 20,000/microliter above baseline at six months or stable platelet counts with transfusion independence, an increase in hemoglobin by > 1.5g/dL or a reduction in the units of PRBC transfusions by at least 50% during the eight consecutive weeks prior to response assessment - compared with the pretreatment transfusion number in the previous 8 weeks; at least a 100% increase in ANC, or an ANC increase >0.5 x 109/L; and >= 2-fold increase in normal marrow CD34+ cells by CD34 immunohistochemistry or flow cytometry, and/or >= 2-fold increase in normal marrow cellularity as measured by standard stains (H&E) of bone marrow biopsy/aspirate sections.
Toxicity profile | 6 months
  Toxicity profile assessed at 6 months using the CTCAE criteria

SECONDARY OUTCOMES:
Toxicities with extended duration of therapy | 3month, 6month (primary endpoint), every 6 month for 3 years after signing the extension part of the protocol
Serum cytokine profile, i.e. TNFalpha, IFNgamma, TPO | At baseline, 3 and 6 months
Relapse | During 3 Years after Treatment
Multicolor flow cytometry of bone marrow cells | At baseline, 3 and 6 months
Impact of treatment and treatment response on quality of life | 3 month and 6 month
Impact of EPAG on other organ systems commonly involved in FA (e.g. skin lesions, endocrine dysfunction, and incidence of new head/neck, oropharyngeal, gastrointestinal, anogenital or skin cancers by clinical assessment) | At baseline, 3 and 6 months
Hematological responses | At 3 Months
Evaluation of global transcriptome in HSPCs (single cell RNA seq) | At baseline and 6 months
Evaluation of DNA repair activity in HSPCs (Gamma H2AX Assay and comet assay) | At baseline, 3 and 6 months
Clonal evolution | 3month, 6month (primary endpoint), every 6 month for 3 years after signing the extension part of the protocol

CONTACTS AND LOCATIONS:
Overall Officials: Andre Larochelle, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-H-0121.html